CLINICAL TRIAL: NCT05639478
Title: Implementing a Contextually Appropriate Intervention Strategy in Primary Care for the Foot-ankle of People With Diabetes to Improve Clinical and Functional Status and Quality of Life
Brief Title: FOot CAre and Exercises ImplementatioN for People With Diabetes in Primary Care
Acronym: FOCAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOCAIN
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Neuropathy, Polyneuropathy (Manifestation)
Keywords: exercise therapy; diabetic foot; preventive care; foot-related exercises; musculoskeletal functions; primary health care
MeSH Terms: conditions — Diabetes Mellitus; Polyneuropathies; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will perform face to face foot-related exercises for 12 weeks.
  Interventions: Other: Foot-related exercises
- Control group (No Intervention): Participants in the control group will not receive any specific intervention in addition to the treatment recommended by the health professionals team (doctors, nurses, podiatrists), which includes pharmacological treatment, and self-care recommendations and foot care by international consensus.

INTERVENTIONS:
Other: Foot-related exercises — Face to face foot-related exercises, supervised by physiotherapist and based in the specific software (Sistema de Orientação do Pé diabético, SOPED) and or booklet, in addition to self-care recommendations and foot care by international consensus. The maximum duration of a session is 40 min and should be be performed 1-2 times/week. The subject should warm-up the foot-ankle and then start exercising in the order suggested by the physiotherapist. The foot exercises progresses from one set with 30 repetitions in a sitting position, to exercising standing, then performing the exercise on one foot only. Other progression criterion is to increase the number of sets performed. The effort scale regulates the individual effort for his/her progression.
  Other Names: Intervention group
  Arms: Intervention group

SUMMARY:
The main objective of this type 2 hybrid implementation effectiveness trial is to implement a contextually appropriate preventive intervention for 12 weeks face to face group foot and ankle exercises for people with diabetic foot in the primary care of the city of Limeira/SP, through the training of Primary Care workers. The study will monitor the implementation itself and the clinical outcomes: clinical and functional status and quality of life.

DETAILED DESCRIPTION:
The study is a type 2 hybrid implementation effectiveness trial, whose objective is to simultaneously test the clinical intervention and the implementation strategy. The study will take place in 4 phases, the first being pre-implementation, whose objective is to gather information about local characteristics, barriers and facilitators, and constitute the implementation team. During the second phase, the implementation team will be responsible for structuring the actions for the implementation of the intervention, adapting it to the context defined in phase 1, developing strategies for the training of primary care workers. In phase 3, we will implement the intervention either using a software or a booklet for people with diabetes and we will monitor the participants' diabetes-related, functional and quality of life outcomes after the 12 weeks of intervention. Reach, adoption and implementation will be evaluated using the RE-AIM tool. In phase 4 - _maintenance - _the municipality will be responsible for maintaining, expanding and improving the changes achieved, promoting the sharing of experience with other public and private institutions, facilitating the diffusion of similar programs. Specifically in the phase 3, a randomized controlled trial will be performed with 356 patients with diabetic neuropathy. The participants will be randomly assigned into either a control group (recommended foot care by international consensus with no foot exercises) or an intervention group that will perform face to face exercises, supervised by physiotherapists for 12-weeks. The subjects will be evaluated in 2 different times to access the effect of the intervention: baseline and 12 weeks, for all outcomes. The following outcomes will be assessed in all times: (1) diabetic neuropathy symptoms by Michigan Neuropathy Screening Instrument, (2) range of motion of the ankle and first metatarsophalangeal joint, (3) fuzzy score of the neuropathy severity, (4) Time up and go, (5) hallux and toes strength (by a pressure plate measurement , (6) hallux strength (by the enhanced paper grip test),(7) ulcers and pre-ulcerative lesions and (8) quality of life (EQ-5D). The hypothesis of this study is that the intervention will reduce the symptoms of diabetic neuropathy, increase the strength of the foot muscles, decrease the severity of the diabetic neuropathy (fuzzy score), decrease the number of neuropathy symptoms, as well increase range of motion, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2;
* Be able to provide consistent information;
* Ability to walk independently for at least 10 meters;
* Availability to participate in the intervention at the established group time.

Exclusion Criteria:

* Neurological and / or rheumatologic diseases diagnosed;
* Perform physiotherapy intervention throughout the intervention period;
* Receiving any physiotherapy intervention or offloading devices;
* Active foot ulcer;
* Major vascular complications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline Diabetic Neuropathy Symptoms at 12-week Instrument | 12 weeks
  Score of the Michigan Neuropathy Screening Instrument (MNSI). This questionnaire comprises 15 questions about symptoms and events related to leg and foot sensitivity and is administered by the participant himself. The answers are summed to get a total score. The sum of all items results in a score ranging from 0 to 13 (13 represents the worst rating of the neuropathy)
Change From Baseline of the Foot and Ankle range of motion at 12-week | 12 weeks
  Ankle and first metatarsophalangeal joint will be measured by manual goniometers.

SECONDARY OUTCOMES:
Change From Baseline of the Fuzzy Classification of the Diabetic Neuropathy Severity at 12-week | 12 weeks
  The fuzzy classification of the diabetic neuropathy severity will be given by the Fuzzy software score developed by the Laboratory of Biomechanics of Movement and Human Posture available free of charge at: http:// www.usp.br/labimph/fuzzy/. It is a decision support system for classification of the diabetic neuropathy. This decision is based on three domains: signs and symptoms extracted from the Michigan Neuropathy Screening Instrument; tactile sensitivity through the number of non-sensible areas using a 10-g monofilament; and vibration sensitivity by vibrating a tuning fork (128Hz) characterized as absent, present or diminished. The software produces a score from 0 to 10 and the higher the score, the more severe the diabetic neuropathy.
Change from baseline of the toes and hallux strength at 12-week | 12 weeks
  Toes and hallux (summed) strength will be measured by a pressure plate with the subjects pressing down the plataform with toes standing.
Change from baseline of the hallux strength at 12-week | 12 weeks
  Hallux strength will be measured by the paper grip test using a card where the examiner places it under the participant's hallux, asking the participant to hold it firmly with the hallux. The examiner pulls the card with increasing force while the participant resists
Change From Baseline Time up and go at 12-week | 12 weeks
  Time spent for the subjects to rise from a standard arm chair, walk to a marker 3 m away, turn, walk back, and sit down again.
Change from baseline of the Quality of life at 12-week | 12 weeks
  Score of the EQ-5D questionnaire answered by the participants, which is a generic instrument for measuring health-related quality of life that allows generating an index representing the value of an individual's health status.
Change From Baseline of the foot ulcers and pre ulcerative lesions at 12-week | 12 weeks
  The presence of ulcers or pre-ulcerative lesions will be monitored through photos without identifying the participant. In cases of doubt, there will be a case discussion with a stoma therapist nurse, specialized in wounds on the feet of people with diabetes
Reach of the implementation at 12-week | 12 weeks
  According to the RE-AIM tool, percentage of coverage and representativeness of people with diabetes participating in the intervention. It will be calculated at the individual level by dividing the population reached by the intervention by the total population of people with diabetes eligible for the intervention. Furthermore, the representativeness of this population will be observed based on sociodemographic data and compared to the non-participating group.
Adoption of the implementation | End of phase 1, end of phase 2
  According to the RE-AIM tool, percentage of coverage and representativeness of locations that we will implement (18 clusters) and key actors participating in phase 1 and in the professional training in phase 2. Representativeness of the participating units and professionals will also be considered in the analysis
Implementation at 12 weeks | 12 weeks
  According to the RE-AIM tool, fidelity to the initially proposed intervention will be evaluated qualitatively and quantitatively, as well as the adaptations - if carried out, through feedback during the course of implementation and in the final evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Isabel CN Sacco, PhD, Study Director — Associate Professor at Medicine of University of São Paulo; Carla BR da Silva, PT, Principal Investigator — Researcher of School of Medicine of University of São Paulo
Locations (1):
- Equipe Multidisciplinar E-Multi, Limeira, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues CB, Soares PNC, Schmitt ACB, Sacco ICN. Implementing a contextually appropriate foot-ankle exercise programme in primary care for the prevention of modifiable risk factors for ulcers in people with diabetes: protocol for a hybrid type 2 study. BMJ Open. 2024 Feb 5;14(2):e078958. doi: 10.1136/bmjopen-2023-078958. PMID 38316587
- See also: University of Sao Paulo website — http://www.usp.br
- See also: Description Laboratory of Biomechanics of Human Movement and Posture website — http://usp.br/labimph